CLINICAL TRIAL: NCT06023056
Title: Influence of Delayed Vaccination of Hepatitis B Vaccine on Vaccination Safety and Immune Response of Newborns After Gastrointestinal Surgery
Brief Title: Hepatitis B Vaccination After Neonatal Surgery
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Hanbin Zhao, Principal Investigator, Children's Hospital of Chongqing Medical University
Other Study IDs: chcmuzhb20221114
Record Dates: First submitted 2022-11-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Vaccination Reaction; Hepatitis B Virus Infection; Digestive System Disorders of Fetus and Newborn; Blood Transfusion Complication; Hepatitis B Vaccine Adverse Reaction
Keywords: Hepatitis B Vaccination Reaction; Hepatitis B Vaccine Adverse Reaction; Neonatal surgery; Gastrointestinal Surgery
MeSH Terms: conditions — Hepatitis B; Transfusion Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Delayed vaccination group after gastrointestinal surgery: Newborns undergoing gastrointestinal surgery are delayed from receiving hepatitis B vaccination in the vaccination institutions due to the impact of surgery.
- The group of vaccination on time after gastrointestinal surgery: Newborns undergoing gastrointestinal surgery shall be vaccinated with hepatitis B vaccine on time by vaccination institutions.
- Control group: Children who are free of disease and have vaccination and physical examination on time.

SUMMARY:
At present, whether the hepatitis B vaccine (HBV) can be vaccinated on time after neonatal surgery has become a common problem for children's families, neonatal surgeons, and vaccination departments, but there are few relevant studies at home and abroad, and there is no corresponding guide or consensus. In the early stage, our research team investigated the vaccination plans of the vaccination units in the main urban areas of Chongqing for such children through telephone follow-up, and found that the practices of each unit were different, all based on their own experience, and there was no clear evidence to support the vaccination or should not be vaccinated, which may cause some children to miss the best vaccination time or increase the risk of vaccination. The center is a relatively large neonatal surgery center in southwest China. The diagnosis and treatment of neonatal digestive tract malformations is at the leading level in China. It can carry out various neonatal operations such as neonatal necrotizing enterocolitis, congenital anorectal malformations, and congenital megacolon. On average, it carries out more than 30 third and fourth grade neonatal gastrointestinal operations every month. It has accumulated a lot of experience in the follow-up of newborns, There is a large amount of clinical data support for children who need to be vaccinated after surgery, so it is planned to follow up the second and third doses of hepatitis B vaccine and whether there are adverse reactions related to vaccination for children who need to be vaccinated after gastrointestinal surgery in the neonatal period, and at the same time check the production of HBsAb after vaccination, The immune response and adverse reactions of hepatitis B vaccine at different time points after surgery were studied to increase clinical evidence for the determination of hepatitis B vaccine vaccination program for newborns after surgery.

DETAILED DESCRIPTION:
Research design

1. Selection of research objects (research population)

Newborns who were screened in the department and met all of the following criteria were included in this study: 1) term infants and the first dose of hepatitis B vaccine had been vaccinated on time; 2) Children with indications for staged gastrointestinal surgery, and the first operation should be performed within 28 days after birth; 3) The child has no immune system disease or serious development defect or dysfunction of heart, brain, liver, kidney and other organs; 4) HBsAg - before initial operation; 5) Prenatal HBsAg - detection of the mother or father of the child; 6) The guardian signed the informed consent form and agreed to participate in the study. Exclusion criteria: 1) premature infants; 2) The first operation time exceeds 28 days after birth; 3) There are serious developmental malformations or dysfunction of heart, brain, liver, kidney and other organs or immune system diseases; 4) The patient or one of his parents is HBsAg+; 5) Children who are allergic to hepatitis B vaccine or have other serious adverse reactions; 6) Children interviewed by vector.

The end point of the study is 6 years after joining the group. Two mid-term evaluations will be conducted one year and two years after the start of the study. This project will apply for funding until the mid-term evaluation of the first year. The follow-up research funds will be supported by the follow-up projects or self raised funds. The criteria for withdrawal from the cohort were: during the study period, the children were infected with hepatitis B virus due to other reasons such as "surgery, blood transfusion, trauma", or diagnosed with immune related diseases during the follow-up period.

2. Patient grouping

1. Newborns who need to undergo gastrointestinal staging surgery as the research object can be included in this study after meeting the inclusion criteria and obtaining the consent of the guardian;
2. The children included in this study were divided into "delayed vaccination group after surgery" and "standard vaccination group after surgery" according to the evaluation of the community vaccination department. At the same time, 1-year-old and 2-year-old children with indirect inguinal hernia who were vaccinated according to the standard immunization program and had no other diseases were taken as the "control group";
3. Collect the general information of the "delayed vaccination group after operation" and the "standard vaccination group after operation", the mother's prenatal hepatitis B two-and-a-half, the children's hepatitis B vaccination time, the adverse reactions of hepatitis B vaccination, and the children's hepatitis B two-and-a-half before each hospitalization operation and at the age of 1 and 2; The level of hepatitis B surface antibody in delayed vaccination group, standard vaccination group and control group was compared;
4. Collect the remaining serum of "Postoperative Delayed Inoculation Group" and "Postoperative Standard Inoculation Group" for HBV DNA detection;
5. The definition of bias refers to ROBINS-I standard, including bias caused by confusion, bias in the selection of research objects, bias in the classification of intervention measures, bias deviating from the expected intervention measures, bias caused by missing data in the outcome measurement and bias in selective reporting of results. Bias is divided into four levels: mild, moderate, severe and extremely severe.

3. Interventions

All the operated children were treated in Liangjiang Neonatal Surgery Department of Children's Hospital Affiliated to Chongqing Medical University. Before operation, they were examined for hepatitis B and HBV DNA.

4. Follow up plan

Collect the general information of the "delayed vaccination group after operation" and the "standard vaccination group after operation", the mother's prenatal hepatitis B two-and-a-half, the children's hepatitis B vaccination time, the adverse reactions of hepatitis B vaccination, and the children's hepatitis B two-and-a-half before each hospitalization operation and at the age of 1 and 2; The level of hepatitis B surface antibody in delayed vaccination group, standard vaccination group and control group was compared; Collect the remaining serum of "Postoperative Delayed Inoculation Group" and "Postoperative Standard Inoculation Group" for HBV DNA detection;

5. Main measurement indexes

Collect the general information of the enrolled children, the mother's two pairs and a half of hepatitis B before delivery, the children's hepatitis B vaccination time, the adverse reactions of hepatitis B vaccination, and the children's two pairs and a half of hepatitis B before each hospitalization operation and at the age of 1 and 2; The level of hepatitis B surface antibody in the delayed vaccination group, the standard vaccination group and the control group were compared.

6. Sample size calculation

According to the previous statistics, the average value of HBsAb of 992 neonates in our outpatient department was 349.5 IU/L, the standard deviation was 420.59 IU/L, and the average value of HBsAb of 1317 1-year-old children was 575.5 IU/L. Therefore, it is estimated that HBsAb will increase by 226 IU/L during the 1-year follow-up α= 0.05， β= 0.1, calculated according to the following formula.

Data management

1. Data entry

   This project uses EpiData to establish the database. The database designer determines the database creation requirements and database structure according to the case report form (CRF form) to ensure that the database content and structure are consistent with the CRF form, and the specified data can be properly entered into the database. The xx database is strictly password protected, and only the personnel directly involved in the research can obtain the password/account. According to the original observation records of the subjects, the researchers timely, completely, correctly and clearly loaded the data into the CRF table. The CRF form reviewed and signed by the investigator shall be submitted to the clinical research data administrator in time. The research data are entered into the EpiData database by authorized researchers. The database system of EpiData is used for double person and double computer input, and then the database is compared twice. Data changes due to input errors or other reasons will be recorded in detail and confirmed by the researcher. The questions and answers between the data administrator and the researcher are in the form of question table, which is kept for future reference.
2. Contents and methods of data verification and management

   Key points and process of data verification, as well as requirements for data locking. For example, when all case report forms have been entered in duplicate and checked without error, data cleaning has been completed, all queries have been answered or explained, and data quality control has been completed, the data administrator will write a database inspection report, which includes the completion of the study (including the list of dropped subjects), inclusion/exclusion criteria, integrity check, logic consistency check, outlier data check, time window check, drug combination check Adverse event inspection, etc. The researcher confirmed that the database will be locked.
3. Safety evaluation

   All adverse events were recorded. In particular, incidents that resulted in hospitalization, prolonged hospitalization, additional surgical or medical treatment, or death were reported.
4. Quality control and quality management

Before the start of the study, patients were enrolled in strict accordance with the inclusion and exclusion criteria, standardized case report forms (CRF) were developed, and ethical review and clinical study registration were confirmed; During the research, ensure the integrity of CRF table data records, the consistency of original data and CRF data, the security of data archiving, review the completion progress and queue interruption, and analyze the preciseness of data; After the study, confirm the integrity of statistical data, the standardization of statistical methods, the standardization of paper writing, and update the clinical study registration data.

ELIGIBILITY:
Inclusion Criteria:

1. Term neonates; 2. Underwent staged gastrointestinal surgery; 3. HBsAg-; 4. No immune system disease; 5.no serious defect of heart, brain, liver, kidney and other organs.

Exclusion Criteria:

1. Premature; 2. HBsAg+; 3. Having immune system diseases; 4. Having serious defect of heart, brain, liver, kidney and other organs; 5. Lost patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Follow up the neonates who live in the medical institution and meet the inclusion criteria. The end point of the study is 6 years after enrollment. Two mid-term evaluations will be conducted one year and two years after the start of the study. This project applies for funding until the mid-term evaluation of the first year. The follow-up research funds will be supported by the follow-up projects or self raised funds. The criteria for withdrawal from the cohort were: during the study period, the children were infected with hepatitis B virus due to other reasons such as "surgery, blood transfusion, trauma", or diagnosed with immune related diseases during the follow-up period.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2030-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Prenatal hepatitis B surface markers | 1 month
  Prenatal hepatitis B surface makers (HBsAg, HBsAb, HBeAg, HBeAb, HBcAb) of mothers and childrens. Measurement of relevant indicators using Roche chemiluminescence method.
Newborn condition | 1 month
  Surface markers of hepatitis B (HBsAg, HBsAb, HBeAg, HBeAb, HBcAb) in newborn.
Vaccination time | up to 2 years
  Time for subjects to receive three doses of hepatitis B vaccine
Adverse reactions | 2 years
  Whether there are vaccine related adverse reactions after vaccination: fever, urticaria, local pain, erythema, induration, atc.
Immune effect of vaccine | up to 2 years
  Results of hepatitis B surface markers (HBsAg, HBsAb, HBeAg, HBeAb, HBcAb) at the age of 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Hanbin Zhao, Doctor, Principal Investigator — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We will decide whether to open the case according to the willingness to finally include the case.

REFERENCES:
- [Background] National Center for Immunization and Respiratory Diseases. General recommendations on immunization --- recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2011 Jan 28;60(2):1-64. PMID 21293327
- [Background] Szilagyi PG, Rodewald LE. Missed opportunities for immunizations: a review of the evidence. J Public Health Manag Pract. 1996 Winter;2(1):18-25. doi: 10.1097/00124784-199600210-00005. PMID 10186652